CLINICAL TRIAL: NCT05751733
Title: Apatinib Mesylate Versus Standard Second-line TKI in the Treatment of Advanced Gastrointestinal Stromal Tumors: a Randomized, Open, Controlled, Single-center Clinical Study
Brief Title: Apatinib Mesylate Versus Standard Second-line TKI in the Treatment of Advanced GIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYGIST202202
Record Dates: First submitted 2023-02-08; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; Apatinib mesylate; tyrosine kinase inhibitors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — apatinib; Sunitinib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Subjects received Apatinib mesylate
  Interventions: Drug: Apatinib Mesylate
- Control group (Active Comparator): Subjects received TKI second-line therapy such as Sunitinib, Imatinib plus, Dasatinib, and Reveratinib.
  Interventions: Drug: Sunitinib, Imatinib dosage, Dasatinib, Reveratinib

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib Mesylate (Etan) is a new type of small molecule anti-angiogenic agent, which is a small molecule TKI against VEGFR2 independently developed in China and has the effect of anti-C-Kit and PDGFR.
  Arms: Experimental group
Drug: Sunitinib, Imatinib dosage, Dasatinib, Reveratinib — Second-line TKI drugs
  Arms: Control group

SUMMARY:
The goal of this Mesylate apatinib versus standard second-line TKI in the treatment of advanced gastrointestinal stromal tumors: a randomized, open, controlled, single-center clinical study is to explore the efficacy and safety of Apatinib compared with second-line treatment in advanced GIST patients with first-line TKI failure. The main questions it aims to answer are:

* To explore the efficacy and safety of Apatinib compared with standard second-line treatment for GIST with advanced first-line TKI failure.
* To explore the expression level and MVD value of VEGFR2 in GIST, and to explore the relationship between the expression level and the location, size, mitotic image and recurrence risk grading of GIST.

Patients with advanced GIST were randomly included in the trial group and the control group at a ratio of 1:1.

DETAILED DESCRIPTION:
The objectives of this study were as follows:

1. To explore the efficacy and safety of Apatinib compared with standard second-line treatment of advanced GIST with first-line TKI failure, and to provide high-level clinical evidence for the treatment of late-stage plasmatoma;
2. Explore the expression level and MVD value of VEGFR2 in GIST, and explore the relationship between the expression level and the location, size, mitotic image and recurrence risk grading of GIST.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were enrolled voluntarily and signed a written informed consent with good compliance and follow-up;
2. Age ≥18 years (calculated on the date of signing the informed consent) for both men and women;
3. Previous first-line TKI (Imatinib/Avatinib) therapy and eventual treatment failure (disease progression or toxicity intolerance during treatment);
4. Subjects who provide pre-C-Kit /PDGFRA test reporting can provide 10ml blood sample and fresh or archived tumor tissue for genetic testing.
5. ECOG score: 0 ~ 1;
6. Predicted survival ≥12 weeks.

Exclusion Criteria:

1. Previous molecular targeted therapy other than imatinib/Avatinib for the treatment of gastrointestinal stromal tumor;
2. Toxicity of previous imatinib/Avatinib treatment or other treatments has not recovered or reached NCICTCAE5.0≤ level 1;
3. Patients with clinical symptoms of ascites or pleural effusion who need puncture drainage or who have received thoracic and ascites drainage within 1 month before signing informed consent, except those who only show a small amount of ascites or pleural effusion without clinical symptoms;
4. A second primary malignancy within the last 5 years, except for basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix that has been adequately treated;
5. Gastrointestinal stromal tumor with central nervous system metastasis;
6. Inability to swallow, chronic diarrhea and intestinal obstruction, with multiple factors affecting drug administration and absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free survival (PFS) | 12 months
  Progression-free survival is the time from treatment to observed disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  Overall Survival is the time from randomization to death from any cause.For subjects who had been lost to follow-up prior to death, the last follow-up time was usually calculated as the time of death.
Objective Response Rate (ORR) | 24 months
  Objective response rate refers to the proportion of patients whose tumor volume has decreased to a predetermined value and can maintain the minimum time limit, including complete response (CR) and partial response (PR) cases.
Disease Control Rate (DCR) | 24 months
  Disease control rate (DCR) refers to the proportion of patients whose tumors shrink or stabilize for a certain period of time, including complete response (CR), partial response (PR), and stable disease (SD) cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided